CLINICAL TRIAL: NCT05376982
Title: Comparison of Neurodevelopmental Treatment Vs Body Weight Supported Treadmill Training Along With Conventional Therapy on Lower Extremity Among Chronic Stroke Patients
Brief Title: Comparison of NT Vs Body Weight Supported TT Along With CT on Lower Extremity in Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall17/506
Record Dates: First submitted 2022-05-05; First posted 2022-05-17 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Chronic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurodevelopmental Treatment (Experimental): Using Neurodevelopmental Treatment Method
  Interventions: Diagnostic Test: Neurodevelopmental Treatment
- Body weight supported treadmill training along with conventional therapy (Experimental): Using Body weight supported treadmill training along with conventional therapy Method
  Interventions: Diagnostic Test: Body weight supported treadmill training along with conventional therapy

INTERVENTIONS:
Diagnostic Test: Neurodevelopmental Treatment — Using Neurodevelopmental Treatment Method
  Arms: Neurodevelopmental Treatment
Diagnostic Test: Body weight supported treadmill training along with conventional therapy — Using Body weight supported treadmill training along with conventional therapy Method
  Arms: Body weight supported treadmill training along with conventional therapy

SUMMARY:
To determine the effect of Neurodevelopment Treatment vs Body Weight Supported Treadmill Training along with conventional therapy on lower extremity among chronic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Application of M-Cog test for checking patients cognition.
* Chronic ischemic stroke patients.
* Both Male and Female Patients.
* Patients of 35 or above years of age.

Exclusion Criteria:

* Patients with history of recurrent stroke.
* Patients with lower limb fractures or dislocations.
* Patients with Peripheral vascular disease
* Patients with skin discoloration or skin ulcers.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
For lower extremity among chronic stroke patients | 6 Months
  comparison of neurodevelopmental treatment vs body weight supported treadmill training along with conventional therapy on lower extremity among chronic stroke patients

CONTACTS AND LOCATIONS:
Locations (1):
- • General Hospital. • Chaudhary Muhammad Akram Teaching and Research Hospital, University of Lahore Teaching Hospital, Shadman Medical Center, Services Hospital, Bahria International Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No